CLINICAL TRIAL: NCT06784557
Title: Gut Microbiota Alteration With Atorvastatin/Ezetimibe Combination in Patients With Atherosclerotic Cardiovascular Disease
Brief Title: Effect of Ezetimibe on Gut Microbiota
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0161
Record Dates: First submitted 2024-12-30; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Atherosclerotic Cardiovascular Disease With Dyslipidemia
MeSH Terms: interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin 40mg (Active Comparator)
  Interventions: Drug: Atorvastatin 40mg
- Atorvastatin 20mg+Ezetimibe 10mg (Experimental)
  Interventions: Drug: Atorvastatin 20mg+Ezetimibe 10mg

INTERVENTIONS:
Drug: Atorvastatin 40mg — High intensity HMG-CoA reductase inhibitor
  Arms: Atorvastatin 40mg
Drug: Atorvastatin 20mg+Ezetimibe 10mg — Moderate intensity HMG-CoA reductase inhibitor plus NPC1L1 antagonist
  Arms: Atorvastatin 20mg+Ezetimibe 10mg

SUMMARY:
Ezetimibe exerts its primary effects by inhibiting intestinal cholesterol absorption through the NPC1L1 protein. Beyond this, its impact on gut microbiota remains an area of interest. Gut microbiota has been implicated in cholesterol metabolism and CVD pathogenesis through metabolic and non-metabolic pathways. Modulating gut microbiota has been explored as a potential strategy to prevent CVDs.

Despite its intestinal mechanism, the influence of ezetimibe on gut microbiota composition has not been thoroughly investigated. Future studies are needed to elucidate its potential interactions with gut microbial communities and their implications for cholesterol metabolism and cardiovascular health.

DETAILED DESCRIPTION:
1. Study Period The clinical trial spans 12 weeks to analyze baseline data and changes after treatment.

   The study starts upon IRB approval, with participant recruitment concluding within 24 months and the entire study wrapping up within 48 months.
2. Study Design This is an investigator-initiated, prospective, single-center, open-label, randomized clinical trial.

   It involves 110 coronary artery disease (CAD) patients in need of lipid-lowering therapy, divided into two groups:

   Experimental Group (n=55): Moderate-intensity statin (Atorvastatin 20 mg) combined with Ezetimibe 10 mg.

   Control Group (n=55): High-intensity statin monotherapy (Atorvastatin 40 mg). Primary Outcome: Changes in gut microbiota composition. Secondary Outcomes: Changes in blood lipid levels and inflammatory biomarkers.
3. Methods 3.1. Screening and Enrollment Participants are screened for eligibility based on inclusion and exclusion criteria.

   After providing informed consent, participants are randomized into two groups (1:1 ratio) using a permuted block randomization method.

   For those on prior statin or Ezetimibe therapy, a 2-week washout period is required before enrollment.

   3.2. Study Medication

   Participants receive their assigned treatment for 12 weeks, with medications administered orally once daily at consistent times, irrespective of meals:

   High-Intensity Statin Group: Atorvastatin 40 mg. Combination Therapy Group: Atorvastatin 20 mg + Ezetimibe 10 mg. 3.3. Follow-Up Baseline data, including demographic details, blood tests, and stool samples, are collected at enrollment.

   After 12 weeks of treatment, follow-up includes clinical evaluations, blood tests, and stool sample collection for post-treatment analysis.
4. Efficacy Evaluation 4.1. Primary Endpoint

Gut Microbiota Analysis:

Stool samples are analyzed using 16S rRNA sequencing.

Statistical tests compare microbiota differences:

Between groups at baseline (T-test or Mann-Whitney test). Pre- and post-treatment within groups (Paired t-test or Wilcoxon test). Intergroup changes over time (ANOVA test). 4.2. Secondary Endpoint Similar statistical methods are applied to assess changes in blood lipid levels and inflammatory biomarkers.

4.3. Subgroup Analysis

Specific subgroups undergo additional analysis:

Subgroup 1: Low-risk CAD patients (10-year ASCVD risk <7.5%). Subgroup 2: Patients with poor response to therapy (LDL >70 mg/dL after 12 weeks).

Subgroup 3: Recurrent CAD patients despite optimal therapy. Subgroup stool samples are analyzed using shotgun metagenomic sequencing for detailed microbial insights.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19 to 80 years old
* Criteria for Diagnosis of Coronary Artery Disease:

Patients diagnosed with coronary artery disease through coronary angiography, or

Patients who require high-intensity lipid-lowering therapy according to current guidelines:

Clinical atherosclerotic cardiovascular disease, LDL cholesterol ≥ 190 mg/dL, LDL 70-189 mg/dL in diabetic patients, 10-year calculated atherosclerotic cardiovascular disease risk ≥ 7.5%

- Voluntary Consent: Individuals who have voluntarily agreed to participate in the study and signed the consent form.

Exclusion Criteria:

* Patients with active liver disease or liver disease with AST/ALT levels elevated more than twice the upper limit of normal.
* Individuals with allergies or hypersensitivity to HMG-CoA reductase inhibitors or ezetimibe.
* Individuals with a history of adverse reactions to HMG-CoA reductase inhibitors or ezetimibe.
* Pregnant, breastfeeding, or women of childbearing potential.
* Organ transplant recipients or individuals scheduled for organ transplantation.
* Patients with active malignant tumors.
* Patients with inflammatory bowel disease.
* Patients with wasting diseases, autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis), or connective tissue diseases (e.g., systemic sclerosis, polymyositis, and dermatomyositis).
* Patients with a history of taking antibiotics, probiotics, or ezetimibe within 3 months prior to study screening.
* Patients who have undergone gastrointestinal surgery within the past year.
* Patients who do not understand the study content or are unable to provide consent.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut Microbiota After 12 Weeks of Treatment | 12 weeks
  Gut Microbiota difference after intervention Stool samples are analyzed using 16S rRNA sequencing.
  Statistical tests compare microbiota differences:
  Between groups at baseline (T-test or Mann-Whitney test). Pre- and post-treatment within groups (Paired t-test or Wilcoxon test). Intergroup changes over time (ANOVA test).

SECONDARY OUTCOMES:
Changes in Blood Lipid Levels and Inflammatory Biomarker Levels After 12 Weeks of Treatment | 12 weeks
  Similar statistical methods are applied to assess changes in blood lipid levels and inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided